CLINICAL TRIAL: NCT06463886
Title: A Randomized Control Trial of Striving Towards EmPowerment and Medication Adherence (STEP-AD)
Brief Title: Striving Towards EmPowerment and Medication Adherence R01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sannisha K Dale, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230854; R01MH135833 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Mental Health Issue
Keywords: HIV; Black women; Trauma; Intersectional; Discrimination; Stigma; Medication adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Wounds and Injuries; Social Stigma; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP-AD (Experimental): Participants in this arm will receive the manualized 10 session behavioral medicine intervention titled "Striving Towards EmPowerment and Medication Adherence". Participants will be in this group for a total of up to 1.5 years.
  Interventions: Behavioral: STEP-AD
- Enhanced treatment as usual (Active Comparator): Participants in the comparison condition will also complete 10 in person sessions. The first session will consist of a session on healthy living with HIV. The remaining 9 sessions will consist of neutral (daily events) writing. Participants will be in this group for a total of up to 1.5 years.
  Interventions: Behavioral: Enhanced treatment as usual (E-TAU)

INTERVENTIONS:
Behavioral: STEP-AD — This in-person STEP-AD intervention will consist of 10 sessions. Session 1: Life Steps Adherence Session 2: Psychoeducation on the treatment model Session 3: Substance Use and Enhancing Resilience Session 4: Trauma Impact Session 5: Cognitive Restructuring Session 6: Racial Discrimination Impact and Coping Session 7: HIV Stigma Impact and Coping Session 8: Gender-related Stressors and Coping Session 9: Body Image and Healthy Relationships Session 10: Practice, Review, and Relapse Prevention. Each session lasts for about 40 to 60 minutes.
  Arms: STEP-AD
Behavioral: Enhanced treatment as usual (E-TAU) — Participants assigned to the E-TAU condition will receive 10 in person sessions to ensure comparable contact time with study staff and identical incentives. The first session will consist of a session on healthy living with HIV (CDC content on HIV 101 [highlights importance of engaging in care, adhering to medication, finding support], nutrition, and physical activity. The remaining 9 sessions will consist of neutral (daily events) writing. Women will be asked to write a description of their plans for the next 24 hours.
  Arms: Enhanced treatment as usual

SUMMARY:
This is a study for Black women living with HIV to test a counseling program for Black women living with HIV. This participant may be a good fit if the participant is a Black woman, living with HIV, has a history of trauma, and is currently taking Antiretroviral Therapy (ART) medicines

ELIGIBILITY:
Inclusion criteria:

1. Black
2. Living with HIV
3. Cis-gender female
4. Age 18 or older
5. English speaking
6. Viral load non-suppression (>200 ml) within the past year or a lack of HIV viral load measure for 6 consecutive months or more during the past 12 months
7. History of trauma/abuse
8. Capable of completing and fully understanding the informed consent process and study procedures

Exclusion criteria:

1. Unable to completely and fully understand the informed consent process and the study procedures
2. Significantly interfering mental health symptoms (e.g., active psychosis that is untreated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in viral suppression | Baseline up to 1.5 years
  HIV viral load <200 copies/ml time averaged. Measured by blood specimen.

SECONDARY OUTCOMES:
Change in antiretroviral (ART) adherence | Baseline up to 1.5 years
  A 3-item self-report instrument that will measure reported adherence to ART. Responses range from 1 to 6. Responses will be averaged (min average of 1, max average of 6) across items with higher scores indicating higher adherence to ART medication.
Change in adherence to anti-retroviral medications questionnaire | Baseline up to 1.5 years
  A list of 12 reasons why individuals may miss taking their ART (e.g., forgot, change in routine) will be used from the AIDS Clinical Trials Group. The minimum score is 0 (no endorsed reasons for missing medication) and maximum score is 36 (endorsing more reasons for missing ART medication).
Change in engagement in HIV care | Baseline up to 1.5 years
  Number of kept versus number of scheduled visits verified by self-report.
Change in PTSD as measured by PCL-5 | Baseline up to 1.5 years
  Measured by the Posttraumatic Stress Disorder Checklist (PCL)-5, a 20-item self-report measure of PTSD symptoms. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores indicate higher PTSD severity.
Change in Post-traumatic cognitions measured by PTCI | Baseline up to 1.5 years
  The Posttraumatic Cognitions Inventory (PTCI) is a 36-item, self-report questionnaire, and each item is rated on a 7-point Likert scale that ranges from 1 (totally agree) to 7 (totally disagree).
Change in Post-traumatic Stress Disorder Diagnosis | Baseline up to 1.5 years
  A structured mental health diagnostic interview will be administered to evaluate participants' mental health symptoms and whether they meet criteria for mental health diagnoses (e.g. Post-traumatic Stress Disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Sannisha Dale, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No